CLINICAL TRIAL: NCT02930135
Title: Evaluation of Post Operative Pain Following Indirect Pulp Treatment in Young Permanent Teeth Using Antibacterial Versus Conventional Two-Step Bonding System: A Randomized Clinical Trial
Brief Title: Evaluation of Post Operative Pain Following Indirect Pulp Capping Using Antibacterial Bonding System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Sabry Mostafa El Hanafy, Assistant Lecturer in Pediatric Dentistry and Dental Public Health Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-2014
Record Dates: First submitted 2016-10-03; First posted 2016-10-12 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Deep Caries
Keywords: Indirect Pulp Capping, Young Permanent Molars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibacterial Bond (Experimental): Indirect pulp capping using antibacterial bond and x-tra fil composite
  1. Local anesthesia administration
  2. Isolation of tooth with rubber dam
  3. Opening of the cavity and the removal of undermined enamel
  4. Caries at the lateral walls of the cavity and at the dentin-enamel junction is completely removed
  5. Partial removal of carious dentin on the pulp wall.
  6. Washing the cavity and dryness
  7. Apply antibacterial light-cure, self-etching bonding agent (Clearfil SE Protect, Kuraray America, Inc.)
  8. Light-cured bulk fill composite (x-tra fil, VOCO) used as final tooth restoration.
  Interventions: Procedure: Indirect pulp capping
- Conventional Bond (Active Comparator): Indirect pulp capping using conventional bond and x-tra fil composite
  1. Local anesthesia administration
  2. Isolation of tooth with rubber dam
  3. Opening of the cavity and the removal of undermined enamel
  4. Caries at the lateral walls of the cavity and at the dentin-enamel junction is completely removed
  5. Partial removal of carious dentin on the pulp wall.
  6. Washing the cavity and dryness
  7. Apply conventional light-cure, self-etching bonding agent (Clearfil SE Bond, Kuraray America, Inc.)
  8. Light-cured bulk fill composite (x-tra fil, VOCO) used as final tooth restoration.
  Interventions: Procedure: Indirect pulp capping

INTERVENTIONS:
Procedure: Indirect pulp capping — Removal of superficial caries in young permanent molars that my expose tooth pulp if totally removed leaving deep carious layers to be sealed inside with two step bonding system and bulk fill composite as a final restoration
  Other Names: Partial caries removal

SUMMARY:
The aim of this study is to compare the clinical and radiographic success of indirect pulp capping of vital young permanent teeth with deep caries using two-step antibacterial bonding system versus conventional one.

DETAILED DESCRIPTION:
The study was carried out on patients attending outpatient clinic in Pediatric and Dental Public Health department- Faculty of Oral and Dental Medicine Cairo University- Egypt.

**Sample size: On searching, no previous studies were conducted using neither conventional bonding nor antibacterial bonding in indirect pulp treatment in young permanent teeth, so sample size will be measured by estimation rather than calculation.

So, all patients attended outpatient clinic in Pediatric and Dental Public Health department- Faculty of Oral and Dental Medicine Cairo University- Egypt, In the period from 1/8/2015 - 31/10/2015 were enrolled for this study if they compatible with eligibility criteria.

**Clinical Procedures:

I. Diagnosis:

Full personal, medical and dental history,clinical and radiographic examination.

II. Allocation concealment:

Selected envelopes will be opened in the first visit to allocate the patients to their treatment groups .

III.Intervention:

A- Experimental Group: Indirect pulp capping with Antibacterial Two-Step Bonding System:

1. Local anesthesia.
2. Isolation of tooth with rubber dam.
3. Opening of the cavity and the removal of undermined enamel using high speed hand-piece with copious air/water spray and round burs.
4. Caries at the lateral walls of the cavity and at the dentin-enamel junction is completely removed with excavators or low speed round burs.
5. Partial removal of carious dentin (only soft disorganized dentin is removed) on the pulp wall.
6. Washing the cavity with distilled water and dryness with triple airway syringe and sterile cotton.
7. Apply antibacterial light-cure, self-etching bonding agent (Clearfil SE Protect, Kuraray America, Inc.)
8. Light-cured bulk fill composite (x-tra fil, VOCO) will be used as final tooth restoration.
9. Postoperative digital radiograph will be taken as a base line.

B- Comparative Group: Indirect pulp capping with Conventional Two-Step Bonding System Same as that of the experimental group EXCEPT steps number 5 as conventional light-cure, self-etching bonding agent (Clearfil SE Bond, Kuraray America, Inc.) will be applied into cavity according to manufacturer's instruction.

IV. Follow up and postoperative instructions:

- Patients will be recalled 48 hours after the treatment then at 2, 9 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients free from any systemic diseases.
2. Young permanent molars with deep carious lesions according to clinical and radiographic examination and at risk of pulp exposure if complete caries is removed.
3. Absence of clinical pathologic signs (fistula, swelling and abnormal tooth mobility)
4. The absence of clinical symptoms of irreversible pulpitis such as spontaneous pain or pain persisting after the disappearance of the existing stimulus or sensitivity to pressure.
5. Absence of adverse radiographic findings (interradicular or periapical radiolucencies, thickening of the periodontal membrane space, internal and external root resorption).
6. Compliant patient/parent.

Exclusion Criteria:

1. Teeth with previous restorative treatment.
2. Unrestorable teeth.
3. Uncooperative patients.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
change/evidence of post treatment spontaneous and provoked pain by questioning the patients | Immediate post operative, 2, 9 month
  The patients are questioned if they experienced post-operative pain within the first 48 hours and then followed up after 2, 6, 9 month to check if there is a change in the situation and evidence of a complain

SECONDARY OUTCOMES:
Absence of pain on percussion | Immediate post operative, 2, 9 month
  Tapping the tooth occlusal surface using dental mirror, parallel to long axis of the tooth. check patient response if there is pain on percussion.
Absence of post treatment swelling | Immediate post operative, 2, 9 month
  Visual inspection of the gingiva, buccal and lingual mucoperiosteum related to the tooth if there is any swelling
Absence of adverse radiographic findings | Immediate post operative, 2, 9 month
  Interradicular or periapical radiolucencies, thickening of the periodontal membrane space, internal and external root resorption

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M Moheb, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miyashita H, Worthington HV, Qualtrough A, Plasschaert A. Pulp management for caries in adults: maintaining pulp vitality. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004484. doi: 10.1002/14651858.CD004484.pub2. PMID 17443547
- [Background] Orhan AI, Oz FT, Ozcelik B, Orhan K. A clinical and microbiological comparative study of deep carious lesion treatment in deciduous and young permanent molars. Clin Oral Investig. 2008 Dec;12(4):369-78. doi: 10.1007/s00784-008-0208-6. Epub 2008 Jun 12. PMID 18548292
- [Background] Maltz M, Garcia R, Jardim JJ, de Paula LM, Yamaguti PM, Moura MS, Garcia F, Nascimento C, Oliveira A, Mestrinho HD. Randomized trial of partial vs. stepwise caries removal: 3-year follow-up. J Dent Res. 2012 Nov;91(11):1026-31. doi: 10.1177/0022034512460403. Epub 2012 Sep 14. PMID 22983407
- [Background] Reichert C. Randomized trial of partial vs. stepwise caries removal: 3-year follow-up. J Orofac Orthop. 2013 May 8. doi: 10.1007/s00056-013-0147-y. Online ahead of print. No abstract available. PMID 23649283
- [Background] Bergenholtz G, Axelsson S, Davidson T, Frisk F, Hakeberg M, Kvist T, Norlund A, Petersson A, Portenier I, Sandberg H, Tranaeus S, Mejare I. Treatment of pulps in teeth affected by deep caries - A systematic review of the literature. Singapore Dent J. 2013 Dec;34(1):1-12. doi: 10.1016/j.sdj.2013.11.001. PMID 24360260